CLINICAL TRIAL: NCT00899054
Title: An Open Label, Multicenter Phase I/II Study Of Selective Cyclin Dependent Kinase Inhibitor P276-00 In Combination With Radiation In Subjects With Recurrent And/Or Locally Advanced Squamous Cell Carcinoma Of Head And Neck
Brief Title: Safety and Efficacy Study of P276-00 in Combination With Radiation in Subjects With Advanced Head and Neck Cancer
Acronym: SPARK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/31/08; P276-00/31/08
Record Dates: First submitted 2009-05-06; First posted 2009-05-12 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — P276-00; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P276-00 plus Radiation (Experimental): P276-00:
  Level 1:100 mg/m2/day x 5 q 3 weeks, level 2:140 mg/m2/day x 5 q 3 weeks, level 3: 185 mg/m2/day x 5 q 3 weeks.
  External beam radiotherapy (EBRT):
  2 Gy per day for 5 days a week for a total radiation dose of 60 Gy over 2 cycles (6 weeks)followed by upto 10 additional Gy if required
  Interventions: Drug: P276-00; Radiation: External beam radiotherapy (EBRT)

INTERVENTIONS:
Drug: P276-00 — P276-00 will be administered at different dose levels: level 1: 100 mg/m2/day dose level 2: 140 mg/m2/day dose level 3: 185 mg/m2/day to be given from day 1 to day 5 every 21 days for 2 cycle. P276-00 will be administered as intravenous infusion in 200 ml 5% Dextrose over 30 min from days 1 to 5 per 21 day cycle for two cycles.
Radiation: External beam radiotherapy (EBRT) — All subjects will receive external beam radiotherapy (EBRT)by using standard conventional fractionation i.e. 2 Gy per day for 5 days a week for a total radiation dose of 60 Gy over 6 weeks followed by upto 10 additional Gy if required.
  Other Names: Radiotherapy

SUMMARY:
The purpose of this study is to identify a dose of P276-00 that can be safely administered along with Radiation and to examine safety and efficacy of the combination in treatment of advanced head and neck cancer.

DETAILED DESCRIPTION:
This is an open label single arm multicenter trial to evaluate safety and efficacy of P276-00 in combination with radiation in patients with recurrent and/or locally advanced squamous cell carcinoma of head and neck. The Primary objective of this study is to determine maximum tolerated dose (MTD) and dose limiting toxicity (ies) (DLT/s) of P276-00 in combination with radiation in subjects with recurrent and/or locally advanced squamous cell carcinoma of head and neck (SCCHN). The Secondary objectives are 1. To evaluate safety and tolerability of the combination regimen of P276-00 and radiation in the study population 2. To analyze pharmacokinetics (PK) of P276-00 in the study population 3. To evaluate efficacy of the combination regimen of P276-00 and radiation in the study population 4. To perform exploratory analysis of biomarkers associated with use of P276-00 and radiation in the study population. In phase 1 component,a cohort of 3 subjects will be enrolled at starting dose level of P276-00 which is 100 mg/m2/day to be given intravenously from day 1 to day 5 in 21 day cycle for 2 cycles in combination with radiation. If this dose is well tolerated then next cohort will be enrolled at higher dose level of P276-00. P276-00 dose escalation will continue until MTD of P276-00 in combination with Radiation is determined. The subsequent dose levels of P276-00 will be 140 mg/m2/day and 185 mg/m2/day.

In phase 2 component 10 subjects will be enrolled at this MTD of P276-00 in combination with radiation to evaluate efficacy. Dose of radiation for both phases is 60 Gy over 6 weeks. Safety evaluations will be conducted at regular intervals during the study. Tumor measurements will be undertaken at baseline, at the end of cycle 2 and 5 to 6 weeks after end of cycle 2. Response evaluation will be performed by Response Evaluation Criteria in Solid Tumors (RECIST). Subjects showing stable disease or better response at the last assessment will be followed up for tumor measurements until progression or recurrence of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Disease specifications:

   * Phase I component: Radiation naïve subjects with histologically and/ or cytologically confirmed squamous cell carcinoma of head and neck that is non-metastatic, unresectable and recurrent. Radiation naïve subjects with non-recurrent, non-metastatic, unresectable, disease can also be enrolled if he/she is intolerant to and/or unwilling for chemoradiotherapy involving standard cytotoxic agents (e.g. cisplatin, carboplatin, oxaliplatin, 5-FU, taxanes, methotrexate, etc)
   * Phase II component: Radiation naïve subjects with non-recurrent, non-metastatic, unresectable, locally advanced squamous cell carcinoma of head and neck who are intolerant to and/or unwilling for chemoradiotherapy involving standard cytotoxic agents (e.g. cisplatin, carboplatin, oxaliplatin, 5-FU, taxanes, methotrexate, etc).
2. Treatment specifications:

   * Phase I Component: subjects must not have received any treatment (chemotherapy, targeted or biologic agents, radiotherapy, surgery etc) for the recurrent disease.
   * Phase II Component: The subjects must not have been curatively operated for the disease.
3. Subjects must have completed any prior chemotherapy, biologic/targeted anti-cancer therapy or surgery at least 4 weeks (at least 6 weeks for nitrosureas and mitomycin C) before initiation of protocol treatment and subjects must have recovered (to < or = grade 1) from the toxic effects from any prior therapy
4. Measurable disease as per RECIST criteria.
5. Age > or = 18 years
6. ECOG (Eastern Cooperative Oncology Group) performance status < or = 2
7. Life expectancy of at least 12 weeks
8. Normal organ and marrow function:

   * Hemoglobin > or = 100 g/L
   * Leukocytes > or = 3 x 109/L
   * Absolute Neutrophil Count (ANC)> or = 1.5 x 109/L
   * Platelets > or = 75 x 109/L
   * Total bilirubin < or = 1.5 X institutional Upper Limit of Normal (ULN)
   * AST(SGOT)< or = 2.5 X institutional ULN
   * ALT(SGPT)< or = 2.5 X institutional ULN
   * Creatinine < or = 1.5 X institutional ULN
9. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Nasopharyngeal carcinoma
2. Subjects who had received any other investigational drug within 1 month prior to day 1 of study drug administration or who have not recovered (to < or = grade 1) from adverse effects of the investigational agent received prior to this period.
3. History of unstable angina or myocardial infarction or stroke within 6 months prior to initiation of protocol treatment.
4. QTcF > 450 msec
5. Subjects with uncontrolled inter-current illness including, but not limited to active infection, symptomatic congestive heart failure, cardiac arrhythmia, psychiatric illness or any condition that would limit compliance with study requirements.
6. Subjects known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B.
7. Women who are pregnant or lactating.
8. Women of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use at least two approved methods of contraception, including at least one barrier method prior to study entry (after signing the informed consent document), during the duration of study participation and for at least 4 weeks after withdrawal from the study drug, unless they are surgically sterilised.
9. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at an unacceptable risk or deems the subject not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicity (ies) (DLT/s) of P276-00 in combination with radiation in subjects with recurrent and/or locally advanced squamous cell carcinoma of head and neck (SCCHN) | 3 weeks

SECONDARY OUTCOMES:
To evaluate safety and tolerability of the combination regimen of P276-00 and radiation in the study population | Every week
To analyze pharmacokinetics (PK) of P276-00 in the study population | Day 2 and Day 5 of Cycle 1
To evaluate efficacy of the combination regimen of P276-00 and radiation in the study population | Every 6 weeks
To perform exploratory analysis of biomarkers associated with use of P276-00 and radiation in the study population | Day 1 and Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Kirushna Kumar, MD, RT, Principal Investigator — Meenakshi Mission Hospital & Research Centre, Madurai, India; Raj Nagarkar, MS, Principal Investigator — Curie Manavata Cancer Center, Nashik, India; Subhashini John, MD, DMRT, Principal Investigator — Christian Medical College, Vellore, India; Balaji Shewalkar, MD, DNB, Principal Investigator — Government Medical College, Aurangabad, India; M. Nagarajan, MD, DNB, Principal Investigator — V. N. Cancer Centre, GKNM Hospital, Coimbatore, India; Naresh Somani, DM, Principal Investigator — Bhagwan Mahawir Cancer Hospital & Research Centre, Jaipur, India
Locations (6):
- India (6):
  - Government Medical College, Aurangabad, Maharashtra
  - Curie Manavata Cancer Center, Nashik, Maharashtra
  - Bhagwan Mahawir Cancer Hospital & Research Centre, Jaipur, Rajasthan
  - V. N. Cancer Centre, GKNM Hospital, Coimbatore, Tamil Nadu
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu